CLINICAL TRIAL: NCT07295275
Title: Safety and Efficacy of Trans-arterial Versus Trans-portal ICG Fluorescence-Guided Laparoscopic Liver Watershed Resection: A Multicenter, Ambispective Cohort Study
Brief Title: Safety and Efficacy of Transarterial ICG Fluorescence-Guided Laparoscopic Anatomical Liver Resection
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiwei Huang, Clinical Professor, West China Hospital
Other Study IDs: JHuang20235
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Liver Cancer
Keywords: Laparoscopic Anatomical Liver Resection; Indocyanine Green Fluorescence; Hepatocellular Carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transarterial ICG Group: Patients who underwent laparoscopic anatomical liver resection guided by superselective transarterial injection of ICG.
  Interventions: Procedure: Laparoscopic Anatomical Liver Resection (guided by transarterial injection of ICG)
- Transportal ICG Group: Patients who underwent laparoscopic anatomical liver resection guided by transportal (portal vein) injection of ICG.

INTERVENTIONS:
Procedure: Laparoscopic Anatomical Liver Resection (guided by transarterial injection of ICG) — Laparoscopic liver resection using ICG fluorescence imaging for tumor and liver segment visualization. Comparison lies in the route of ICG administration (Arterial vs. Portal).
  Groups: Transarterial ICG Group

SUMMARY:
This multicenter, ambispective cohort study evaluates the safety and efficacy of trans-arterial Indocyanine Green (ICG) fluorescence-guided laparoscopic liver watershed resection for Hepatocellular Carcinoma (HCC). The study aims to compare the outcomes of the trans-arterial ICG staining approach versus the conventional trans-portal (portal vein) ICG staining approach.

DETAILED DESCRIPTION:
The study employs an ambispective design, comprising:

A Retrospective Cohort: Collecting clinical data from patients treated between June 2020 and August 2025.

A Prospective Cohort: Enrolling new patients from January 2026 to January 2027. Data will be collected from three medical centers. The primary objective is to compare the oncological prognosis, specifically Recurrence-Free Survival (RFS), between the two navigation methods. Secondary objectives include perioperative safety, liver function recovery, and Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Postoperative histopathological diagnosis of Hepatocellular Carcinoma (HCC).
3. Underwent ICG fluorescence-guided laparoscopic anatomical liver resection.
4. Child-Pugh Class A or B.
5. ASA score I-III.
6. ECOG Performance Status 0-2.
7. No invasion of major vessels (main portal vein/first-order branches, main hepatic vein).
8. No distant metastasis.

Exclusion Criteria:

1. Pathology confirms non-HCC components (e.g., cholangiocarcinoma, combined HCC-ICC) or metastatic liver cancer.
2. Concomitant other active malignancies.
3. Preoperative anti-tumor therapy (TACE, ablation, radiotherapy, systemic therapy) or history of prior hepatectomy.
4. Ruptured tumor.
5. Conversion to open surgery.
6. Unclear surgical records regarding ICG staining method.
7. Intraoperative ICG staining failure (e.g., diffuse staining, unclear boundaries) preventing fluorescence-guided resection.
8. Missing data preventing primary endpoint assessment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 80 years with a histopathological diagnosis of Hepatocellular Carcinoma (HCC). The population consists of patients who have undergone (retrospective cohort) or are scheduled to undergo (prospective cohort) laparoscopic anatomical liver resection guided by Indocyanine Green (ICG) fluorescence imaging at one of the participating centers. Participants must have Child-Pugh class A or B liver function and no evidence of major vascular invasion or distant metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to 18 months post-surgery (assessing the 18-month RFS rate as a key benchmark)
  RFS is defined as the time interval from the date of surgery to the date of first documented tumor recurrence (intrahepatic or extrahepatic) or death from any cause. Evaluated using Kaplan-Meier analysis.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 3 years post-surgery
  OS is defined as the time from the date of surgery to the date of death from any cause.
Incidence of Perioperative Complications | From surgery up to 90 days post-surgery
  Number of participants with postoperative complications (e.g., bile leakage, hemorrhage, infection, liver failure), graded according to the Clavien-Dindo classification system.

OTHER OUTCOMES:
Liver Function Recovery | Pre-operative, Post-operative Days 1, 3, 5, and 1 month
  Assessment of dynamic changes in liver function indicators, including Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), and Total Bilirubin (TBIL) levels.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No